CLINICAL TRIAL: NCT06287827
Title: Evaluation of the Treatment of Moderate and Severe Acute Malnutrition in Outpatient Care Services in Venezuela: a Multicentric and Prospective Cohort Research
Brief Title: Treatment of Acute Malnutrition in Outpatient Care Services in Venezuela: a Prospective Cohort Research
Status: Completed | Type: Observational
Sponsor: UNICEF - Venezuela (Other)
Responsible Party: Sponsor
Other Study IDs: 190224
Record Dates: First submitted 2024-02-19; First posted 2024-03-01 (Actual); Last update posted 2024-10-02 (Actual); Status verified 2024-09

CONDITIONS: Acute Malnutrition in Childhood; Wasting; Child Malnutrition
Keywords: Severe acute malnutrition; Moderate acute malnutrition; Ready-to-use therapeutic food; Malnutrition treatment; Venezuela; Mid-upper arm circumference; Wasting; Simplified protocol; Standard protocol
MeSH Terms: conditions — Cachexia; Child Nutrition Disorders; Severe Acute Malnutrition | interventions — AIEOP acute lymphoblastic leukemia protocol

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Simplified protocol: The first cohort will be composed of all children between 6 and 59 months of age who attend predefined outpatient care points in the states Distrito Capital, Miranda, and La Guaira. These children must meet the inclusion criteria for the research. For those selected in these centers, the method of nutritional treatment for acute malnutrition will be the simplified protocol. Adaptations in this protocol include:
  1. Use of a single treatment product (Ready to use therapeutic food).
  2. Reduced dose.
  3. Expanded cut-offs.
  Interventions: Procedure: Simplified protocol
- Standard protocol: The second cohort will be composed of all children between 6 and 59 months of age who attend other predefined outpatient care points in the four states and met the inclusion criteria for this research. Nutritional treatment will be administered to these children, following the WHO Standard Protocol.
  Interventions: Procedure: Standard protocol

INTERVENTIONS:
Procedure: Simplified protocol — MUAC-based dosing:
  * SAM [MUAC <115mm or WHZ <-3 or oedema (+/++)] = Two 92g sachets Ready to use Therapeutic Food (RUTF)/day (Approx. 1000 kcal/day).
  * MAM [MUAC 115mm<125mm or WHZ <-2] = One 92g sachet RUTF/day (Approx. 500 kcal/day).
  Groups: Simplified protocol
Procedure: Standard protocol — Weight-based dosing
  * SAM: Mid-upper-arm circumference (MUAC) <115mm or Weight-Height/length Z Score <-3 or mild or moderate bipedal oedema: 150-185 kcal/kg/day is offered using RUTF until the patient passes to MAM and then the dose is reduced to 100 -130 kcal/kg/day using RUTF until recovery.
  * MAM: MUAC 115-<125mm or Weight-Height/length Z Score <-2: 100-130 kcal/kg/day is offered using RUTF until recovery.
  Groups: Standard protocol

SUMMARY:
The goal of this observational study is to compare the effectiveness, safety, and efficiency of the simplified protocol, which includes the following three modifications: a) use of a single treatment product (RUTF), b) reduced dose, c) expanded cut-offs, with the standard protocol based on the 2023 World Health Organization (WHO) guidelines for the prevention and treatment of acute malnutrition in children aged 6 to 59 months, in outpatient care services of the states of Bolívar, Capital District, La Guaira, and Miranda of Venezuela.

The main question it aims to answer is:

What is the effectiveness, safety, and efficiency of the simplified protocol, which includes these three modifications (use of a single treatment product (RUTF), reduced dose, expanded cut-offs) when compared to a standard protocol that is based on the 2023 WHO guidelines for the prevention and treatment of acute malnutrition in children aged 6 to 59 months in the outpatient care services of the states of Bolívar, Capital District, La Guaira, and Miranda of Venezuela? This prospective cohort, longitudinal study will be conducted in 4 states, treating children aged 6-59 months diagnosed with uncomplicated AM, defined as WHZ <-2 or mid-upper-arm circumference (MUAC) <125mm or bilateral edema. Children will be prospectively followed for 16 weeks or until their recovery.

Researchers will compare the simplified protocol cohort with the standard protocol cohort to determine which one has the best effectiveness, safety, and efficiency indicators in the Venezuela context.

The effectiveness of the treatment will be measured by the recovery rate, duration of the treatment, and changes in anthropometry (weight, height, and arm circumference). Other treatment effects will also be measured, including how many are admitted to the hospital, death, and relapse rates from the nutritional program. An economic evaluation component will be incorporated. Total costs will be aggregated and presented as costs per child treated and per child recovered.

DETAILED DESCRIPTION:
The general objective of the study is to compare the effectiveness, safety, and efficiency of the simplified protocol, which includes the following three modifications: a) use of a single treatment product (RUTF), b) reduced dose, c) expanded cut-offs, with the standard protocol based on the 2023 WHO guidelines for the prevention and treatment of acute malnutrition in children aged 6 to 59 months in outpatient care services in the states Bolívar, Capital District, La Guaira, and Miranda of Venezuela.

This will be a multicentric and prospective cohort study assessing the Simplified Protocol with the Standard Protocol, among children with uncomplicated acute malnutrition. Children will be prospectively followed until their recovery or for a maximum of 16 weeks.

The study will be implemented in 4 Venezuelan states chosen based on their acute malnutrition prevalence and operational constraints.

The protocol will be implemented by health professionals from each institution, duly previously trained in applying the study protocol.

ELIGIBILITY:
Inclusion Criteria:

* Simplified protocol cohort

  * MUAC <125 mm or
  * Weight-Height/length Z Score <-2 or
  * Mild bipedal pitting oedema.

And all the following:

* No medical complications
* Positive appetite test.

  * Standard protocol cohort

SAM:

* MUAC <115 mm or
* Weight-Height/length Z Score <-3 or
* Mild bipedal pitting oedema

And all the following:

* No medical complications
* Positive appetite test

MAM (Although MAM cases are not traditionally included, in this study they will be incorporated if they meet the following criteria):

* MUAC ≥ 115 mm to < 125 mm or
* Weight-Height/length Z Score ≥ -3 to < -2 and
* No nutritional oedema

And at least one the following:

* Failing to recover from moderate wasting after receiving other interventions (counselling alone).
* Having relapsed to moderate wasting
* History of severe wasting
* Households' low socioeconomic status (Determined by Graffar-Mendez-Castellanos method)
* Co-morbidity (HIV, tuberculosis, or a physical or mental disability that does not jeopardize the anthropometric measurements)

Exclusion Criteria:

* Both cohorts:

  * Congenital malformations that make anthropometric measurements impossible.
  * Family that intends to leave the study area before four months.
  * Presence of medical condition requiring referral for hospitalization. Presence of medical condition requiring referral for hospitalization.

Ages: 6 Months to 59 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: The research population consisted of children with uncomplicated moderate or severe acute malnutrition who are admitted to the nutritional care program in care centers and associated institutions in Bolívar, Capital District, La Guaira, and Miranda.
  Given the observational nature of the research, the sample size of the population will not be calculated. Rather, a research group or intentional sample will be analyzed, made up of all children who attend the care centers and meet the inclusion criteria of the research during a collection period of two months in each cohort.
Sampling Method: Non-Probability Sample
Enrollment: 299 (Actual)
Dates: Start 2024-02-14 (Actual); Primary Completion 2024-08-31 (Actual); Study Completion 2024-08-31 (Actual)

PRIMARY OUTCOMES:
Recovery rate | From date of inclusion in the program until the date of recovery or 16th week after inclusion in the program or date of death from any cause, whichever came first
  This indicator is defined as the number of children who recovered from SAM and MAM (WHZ>-2 and MUAC>=125mm and the absence of bilateral edema for two consecutive visits, within 16 weeks of enrollment in the program, divided by the total number of treated children.
Weight gain | From date of inclusion in the program until the date of recovery or 16th week after inclusion in the program or date of death from any cause, whichever came first
  Average weight change in each protocol.
Mid-Upper Arm Circumference (MUAC) gain | From date of inclusion in the program until the date of recovery or 16th week after inclusion in the program or date of death from any cause, whichever came first
  Average Mid-Upper Arm Circumference (MUAC) change in each protocol.
Duration of the treatment | From date of inclusion in the program until the date of recovery or 16th week after inclusion in the program or date of death from any cause, whichever came first
  Defined as the average number of weeks spent on treatment (enrollment and recovery) in children 6-59 months of age at enrollment, according to health registers
Prevalence of child morbidity | From date of enrolment until the date of recovery, last documented progression or date of death from any cause, whichever came first.
  Defined by the number of days with symptoms of acute respiratory infections, fever, diarrhea (three or more loose or liquid stools per day) and malaria divided by the total number of days observed/reported in the recall period
Number of RUTF delivered per child | From date of inclusion in the program until the date of recovery or 16th week after inclusion in the program or date of death from any cause, whichever came first
  Average number of RUTF delivered per child (SAM/MAM) in each protocol
Cost per child | From date of inclusion in the program until the date of recovery or 16th week after inclusion in the program or date of death from any cause, whichever came first
  Average number of dollars that cost to recovery a child in each cohort

SECONDARY OUTCOMES:
Prevalence of child stunting | At the date of recovery or 16th week after inclusion in the program or date of death from any cause, whichever came first
  Proportion of children with Height-for-age Z-score (LAZ)<-2 (according to the 2006 World Health Organization reference) at the end of the study

CONTACTS AND LOCATIONS:
Overall Officials: Pablo Hernandez, MSc, Principal Investigator — Nutri Consult
Locations (4):
- Venezuela (4):
  - Bolivar State Centers, Puerto Ordaz and San Felix, Bolívar
  - Ditrict Capital centers, Caracas, Distrito Federal
  - Miranda State Centers, Santa Lucía, Miranda
  - La Guaira State Centers, La Guaira

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Alvarez Moran JL, Ale GBF, Charle P, Sessions N, Doumbia S, Guerrero S. The effectiveness of treatment for Severe Acute Malnutrition (SAM) delivered by community health workers compared to a traditional facility based model. BMC Health Serv Res. 2018 Mar 27;18(1):207. doi: 10.1186/s12913-018-2987-z. PMID 29580238
- [Background] Bahwere P. Severe acute malnutrition during emergencies: burden management, and gaps. Food Nutr Bull. 2014 Jun;35(2 Suppl):S47-51. doi: 10.1177/15648265140352S107. PMID 25069293
- [Background] Maust A, Koroma AS, Abla C, Molokwu N, Ryan KN, Singh L, Manary MJ. Severe and Moderate Acute Malnutrition Can Be Successfully Managed with an Integrated Protocol in Sierra Leone. J Nutr. 2015 Nov;145(11):2604-9. doi: 10.3945/jn.115.214957. Epub 2015 Sep 30. PMID 26423737
- [Result] Bailey J, Opondo C, Lelijveld N, Marron B, Onyo P, Musyoki EN, Adongo SW, Manary M, Briend A, Kerac M. A simplified, combined protocol versus standard treatment for acute malnutrition in children 6-59 months (ComPAS trial): A cluster-randomized controlled non-inferiority trial in Kenya and South Sudan. PLoS Med. 2020 Jul 9;17(7):e1003192. doi: 10.1371/journal.pmed.1003192. eCollection 2020 Jul. PMID 32645109
- [Result] Stephenson KB, Agapova SE, Hendrixson DT, Koroma AS, Manary MJ. An Optimized Dose of Therapeutic Feeding Results in Noninferior Growth in Midupper Arm Circumference Compared with a Standard Dose in Children in Sierra Leone Recovering from Acute Malnutrition. Curr Dev Nutr. 2021 Feb 2;5(2):nzab007. doi: 10.1093/cdn/nzab007. eCollection 2021 Feb. PMID 33659773
- [Result] James PT, Van den Briel N, Rozet A, Israel AD, Fenn B, Navarro-Colorado C. Low-dose RUTF protocol and improved service delivery lead to good programme outcomes in the treatment of uncomplicated SAM: a programme report from Myanmar. Matern Child Nutr. 2015 Oct;11(4):859-69. doi: 10.1111/mcn.12192. Epub 2015 Apr 7. PMID 25850698
- [Result] Daures M, Phelan K, Issoufou M, Kouanda S, Sawadogo O, Issaley K, Cazes C, Seri B, Ouaro B, Akpakpo B, Mendiboure V, Shepherd S, Becquet R. New approach to simplifying and optimising acute malnutrition treatment in children aged 6-59 months: the OptiMA single-arm proof-of-concept trial in Burkina Faso. Br J Nutr. 2020 Apr 14;123(7):756-767. doi: 10.1017/S0007114519003258. Epub 2019 Dec 10. PMID 31818335
- [Result] Hussain I, Habib A, Ariff S, Khan GN, Rizvi A, Channar S, Hussain A, Fazal S, Kumar D, Alvarez JL, Guerrero S, Grant A, Soofi SB. Effectiveness of management of severe acute malnutrition (SAM) through community health workers as compared to a traditional facility-based model: a cluster randomized controlled trial. Eur J Nutr. 2021 Oct;60(7):3853-3860. doi: 10.1007/s00394-021-02550-y. Epub 2021 Apr 20. PMID 33880645
- [Result] Lelijveld N, Bailey J, Mayberry A, Trenouth L, N'Diaye DS, Haghparast-Bidgoli H, Puett C. The "ComPAS Trial" combined treatment model for acute malnutrition: study protocol for the economic evaluation. Trials. 2018 Apr 24;19(1):252. doi: 10.1186/s13063-018-2594-7. PMID 29690899
- [Result] Bailey J, Lelijveld N, Marron B, Onyoo P, Ho LS, Manary M, Briend A, Opondo C, Kerac M. Combined Protocol for Acute Malnutrition Study (ComPAS) in rural South Sudan and urban Kenya: study protocol for a randomized controlled trial. Trials. 2018 Apr 24;19(1):251. doi: 10.1186/s13063-018-2643-2. PMID 29690916